CLINICAL TRIAL: NCT01120379
Title: XIENCE V® Everolimus Eluting Coronary Stent System (EECSS) USA Post-Approval Study (XIENCE V® USA Long Term Follow-up Cohort)
Brief Title: XIENCE V® Everolimus Eluting Coronary Stent System USA Post-Approval Study (XIENCE V® USA Long Term Follow-up Cohort)
Acronym: XVU-LTF
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-374B
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Coronary Occlusion; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; Stents; Angioplasty; Stent thrombosis
MeSH Terms: conditions — Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- XV-LTF cohort
  Interventions: Device: XIENCE V® EECSS

INTERVENTIONS:
Device: XIENCE V® EECSS — Single-arm study designed to evaluate XIENCE V® EECSS continued safety and effectiveness during commercial use in real world settings.

SUMMARY:
XIENCE V USA is a prospective, multi-center, multi-cohort post-approval study. The objectives of this study are

* To evaluate XIENCE V EECSS continued safety and effectiveness during commercial use in real world settings, and
* To support the Food and Drug Administration (FDA) dual antiplatelet therapy (DAPT) initiative. This initiative is designed to evaluate the composite of all death, myocardial infarction (MI) and stroke (MACCE) and the survival of patients that are free from Academic Research Consortium (ARC) definite or probable stent thrombosis (ST) and that have been treated with drug eluting stents (DES) and extended dual antiplatelet therapy.

DETAILED DESCRIPTION:
Among patients enrolled in the XIENCE V USA who have completed Study Phase I, some will be eligible to participate in the XIENCE V USA Long Term Follow-up (LTF) Cohort. This LTF cohort is a prospective, open-label, multi-center, observational, single-arm study is designed to evaluate XIENCE V EECSS continued safety and effectiveness in real world settings from 1 year after the index procedure up to 5 years. The XIENCE V USA LTF cohort will consist of the following from the initial 5,000 patients:

* The first 1,500 on-label patients who are treated in accordance with the XIENCE V EECSS Instruction for Use (IFU), and consecutively enrolled in the XIENCE V USA study
* The remaining patients who do not participate in the HCRI-DAPT cohort
* Data monitoring committee up to two years

ELIGIBILITY:
Inclusion Criteria:

* The patient agrees to participate in this study by signing the Institutional Review Board approved informed consent form.

Exclusion Criteria:

* The inability to obtain an informed consent.
* Age limit is determined by investigator.
* There are no angiographic inclusion or exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who agree to participate by signing the Institutional Review Board (IRB) approved informed consent form, and who recieve only XIENCE V® EECSS during the index procedure.
Sampling Method: Non-Probability Sample
Enrollment: 5034 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Hermiller, MD, Principal Investigator — Heart Center of Indianapolis; Mitch Krucoff, MD, Principal Investigator — Duke University
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

REFERENCES:
- See also: NCT00676520 — http://www.clinicaltrials.gov/ct2/show/NCT00676520?term=xience+v+usa&rank=3
- See also: NCT01106534 — http://www.clinicaltrials.gov/ct2/show/NCT01106534?term=xience+v+usa&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are derived from the USA interventional cardiology population.
Pre-assignment Details: 8000 patients (5034 patients in initial enrollment phase and 2998 patients in second enrollment phase) were enrolled in XIENCE V USA trial. Out of these 5034 patients, 14 patients were transferred to the HCRI DAPT cohort, leaving 5020 in the XIENCE V USA LTF cohort.
Groups:
- XV-LTF Cohort: XIENCE V® EECSS : Single-arm study designed to evaluate XIENCE V® EECSS continued safety and effectiveness during commercial use in real world settings.
Period: One Year Timepoint
Arm/Group | XV-LTF Cohort
Started | 5020
Completed | 4742
Not Completed | 278
Not completed — Withdrawal by Subject | 41
Not completed — Lost to Follow-up | 115
Not completed — Death | 108
Not completed — Physician Decision | 9
Not completed — Any other reason for early termination | 5
Period: Two Year Timepoint
Arm/Group | XV-LTF Cohort
Started | 4742
Completed | 4505
Not Completed | 237
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 87
Not completed — Death | 123
Not completed — Physician Decision | 12
Not completed — Any other reason for early termination | 4
Period: Three Year Timepoint
Arm/Group | XV-LTF Cohort
Started | 4505
Completed | 4291
Not Completed | 214
Not completed — Withdrawal by Subject | 25
Not completed — Lost to Follow-up | 43
Not completed — Death | 120
Not completed — Physician Decision | 9
Not completed — Any other reason for early termination | 17
Period: Four Year Timepoint
Arm/Group | XV-LTF Cohort
Started | 4291
Completed | 3923
Not Completed | 368
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 10
Not completed — Death | 131
Not completed — Physician Decision | 5
Not completed — Any other reason for early termination | 217

BASELINE CHARACTERISTICS:
Population: Baseline data was analyzed for 5020 patients as out of the enrolled 5034 patients 14 patients were transferred to the HCRI DAPT cohort, leaving 5020 in the XIENCE V USA LTF cohort.
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 5020
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2525
  >=65 years | 2495
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.75 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1564
  Male | 3456
Region of Enrollment [Number; unit: participants]
  United States | 5020

OUTCOME MEASURES:

1. Primary Outcome: Stent Thrombosis (Definite and Probable) Rate as Defined by ARC (Academic Research Consortium)
Description: Stent thrombosis was defined by ARC criteria as definite (angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy), probable (any unexplained death within the first 30 days or, regardless of the time after the index procedure, any MI related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause), and possible (any unexplained death from 30 days after intracoronary stenting until end of trial follow-up). Stent thrombosis was categorized as acute (0-24 hours post stent implantation), subacute (>24 hours to 30 days post stent implantation), late (>30 days to 1 year post stent implantation), or very late (>1 year post stent implantation).
Time Frame: 2 years
Population: Number of participants analyzed excludes patients who are truly lost-to-follow-up, defined as patients who are lost to follow-up through given timepoint without any ARC Defined Patient-Oriented Endpoint (all death, all MI, all revascularization, respectively). Number of participants analyzed includes patients with valid data at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4587
percentage of participants | 1.05 [0.77 to 1.39]

2. Primary Outcome: Stent Thrombosis (Definite and Probable) Rate as Defined by ARC (Academic Research Consortium)
Description: as for outcome 1
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4475
percentage of participants | 1.18 [0.89 to 1.55]

3. Primary Outcome: Stent Thrombosis (Definite and Probable) as Defined by ARC
Description: as for outcome 1
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4093
percentage of participants | 1.56 [1.21 to 1.99]

4. Primary Outcome: Composite Rate of Cardiac Death and Any Myocardial Infarction [MI] (ARC Defined).
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 9.5 [8.64 to 10.32]

5. Primary Outcome: Composite Rate of Cardiac Death and Any Myocardial Infarction (ARC Defined).
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 11.7 [10.78 to 12.63]

6. Primary Outcome: Composite Rate of Cardiac Death and Any Myocardial Infarction (ARC Defined).
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 14.9 [13.90 to 15.99]

7. Secondary Outcome: Composite Rate of All Death and Any MI (Q-wave and Non Q-wave)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 11.8 [10.90 to 12.76]

8. Secondary Outcome: Composite Rate of All Death and Any MI (Q-wave and Non Q-wave)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 15.0 [14.03 to 16.09]

9. Secondary Outcome: Composite Rate of All Death and Any MI (Q-wave and Non Q-wave)
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 19.8 [18.65 to 20.99]

10. Secondary Outcome: Composite Rate of All Death, Any MI (Q-wave and Non Q-wave) and Any Repeat Revascularization (Percutaneous Coronary Intervention [PCI] and Coronary Artery Bypass Graft [CABG]
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 22.4 [21.20 to 23.58]

11. Secondary Outcome: Composite Rate of All Death, Any MI (Q-wave and Non Q-wave) and Any Repeat Revascularization (Percutaneous Coronary Intervention [PCI] and Coronary Artery Bypass Graft [CABG]
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 27.5 [26.20 to 28.76]

12. Secondary Outcome: Composite Rate of All Death, Any MI (Q-wave and Non Q-wave) and Any Repeat Revascularization (Percutaneous Coronary Intervention [PCI] and Coronary Artery Bypass Graft [CABG]
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 34.5 [33.14 to 35.93]

13. Secondary Outcome: Composite Rate of Cardiac Death, Any MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Target Lesion Revascularization (TLR) (PCI and CABG)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 13.3 [12.34 to 14.29]

14. Secondary Outcome: Composite Rate of Cardiac Death, Any MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Target Lesion Revascularization (TLR) (PCI and CABG)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 16.0 [14.96 to 17.06]

15. Secondary Outcome: Composite Rate of Cardiac Death, Any MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Target Lesion Revascularization (TLR) (PCI and CABG)
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 19.7 [18.56 to 20.90]

16. Secondary Outcome: Composite Rate of Cardiac Death and MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Clinically-indicated Target Lesion Revascularization (CI-TLR) (PCI and CABG) (This Composite Endpoint is Also Denoted as TLF)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 13.0 [12.06 to 13.99]

17. Secondary Outcome: Composite Rate of Cardiac Death and MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Clinically-indicated Target Lesion Revascularization (CI-TLR) (PCI and CABG) (This Composite Endpoint is Also Denoted as TLF)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 15.7 [14.65 to 16.74]

18. Secondary Outcome: Composite Rate of Cardiac Death and MI (Q-wave and Non Q-wave) Attributed to the Target Vessel, and Clinically-indicated Target Lesion Revascularization (CI-TLR) (PCI and CABG) (This Composite Endpoint is Also Denoted as TLF)
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 19.3 [18.18 to 20.50]

19. Secondary Outcome: Death (Cardiac Death, Vascular Death, and Non-cardiovascular Death)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 5.4 [4.78 to 6.09]

20. Secondary Outcome: Death (Cardiac Death, Vascular Death, and Non-cardiovascular Death)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 7.6 [6.86 to 8.38]

21. Secondary Outcome: Death (Cardiac Death, Vascular Death, and Non-cardiovascular Death)
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 10.9 [10.01 to 11.85]

22. Secondary Outcome: Any MI (Q-wave and Non Q-wave)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 7.6 [6.85 to 8.38]

23. Secondary Outcome: Any MI (Q-wave and Non Q-wave)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 9.1 [8.29 to 9.95]

24. Secondary Outcome: Any MI (Q-wave and Non Q-wave)
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 11.3 [10.37 to 12.24]

25. Secondary Outcome: Revascularization (Target Lesion, Target Vessel [TVR], and Non-target Vessel) (PCI and CABG)
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4769
percentage of participants | 14.7 [13.69 to 15.71]

26. Secondary Outcome: Revascularization (Target Lesion, Target Vessel [TVR], and Non-target Vessel) (PCI and CABG)
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4741
percentage of participants | 18.2 [17.11 to 19.33]

27. Secondary Outcome: Revascularization (Target Lesion, Target Vessel [TVR], and Non-target Vessel) (PCI and CABG)
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4530
percentage of participants | 22.5 [21.33 to 23.78]

28. Secondary Outcome: Major Bleeding Complications
Description: Major bleeding complications consisted of Clinical Events Committee (CEC)-adjudicated Thrombolysis In Myocardial Infarction (TIMI) major bleeding through 2-year follow-up and site reported major bleeding after 2 years.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4541
percentage of participants | 4.3 [3.68 to 4.88]

29. Secondary Outcome: Major Bleeding Complications (Site Reported)
Description: Major bleeding complications consisted of CEC-adjudicated TIMI major bleeding through 2-year follow-up and site reported major bleeding after 2 years.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4435
percentage of participants | 7.3 [6.56 to 8.11]

30. Secondary Outcome: Major Bleeding Complications
Description: as for outcome 29
Time Frame: 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 4050
percentage of participants | 8.4 [7.54 to 9.27]

31. Secondary Outcome: Dual Antiplatelet Medication Usage
Description: Patient is included if medications (both aspirin and thienopyridine) were taken for at least 1 day during the visit window. The visit window for 2-year visit is 688-772 days.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 5020
percentage of participants | 61.9

32. Secondary Outcome: Dual Antiplatelet Medication Usage
Description: Patient is included if medications (both aspirin and thienopyridine) were taken for at least 1 day during the visit window. The visit window for 3-year visit is 1053-1137 days.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 5020
percentage of participants | 53.1

33. Secondary Outcome: Dual Antiplatelet Medication Usage
Description: Patient is included if medications (both aspirin and thienopyridine) were taken for at least 1 day during the visit window. The visit window for 4-year visit is 1502 days.
Time Frame: 4 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | XV-LTF Cohort
Number analyzed (Participants) | 5020
percentage of participants | 42.5

ADVERSE EVENTS:
Time Frame: Four year endpoint (up to 1502 days)
Description: The number of participants at risk excludes subjects who were early terminated up to 1460 days and had no events through given timepoint.
Arm/Group | XV-LTF Cohort
Serious Adverse Events (participants affected / at risk) | 2730/4852
Other Adverse Events (participants affected / at risk) | 883/4852
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XV-LTF Cohort (N=4852)
Acute coronary syndrome (Cardiac disorders) | 23 (24)
Acute myocardial infarction (Cardiac disorders) | 229 (251)
Angina pectoris (Cardiac disorders) | 784 (1131)
Angina unstable (Cardiac disorders) | 218 (277)
Aortic valve disease (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 22 (22)
Arrhythmia (Cardiac disorders) | 11 (11)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4)
Arteriospasm coronary (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 110 (141)
Atrial flutter (Cardiac disorders) | 37 (47)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 4 (4)
Atrioventricular block complete (Cardiac disorders) | 6 (6)
Atrioventricular block second degree (Cardiac disorders) | 3 (4)
Bradycardia (Cardiac disorders) | 34 (35)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 38 (38)
Cardiac disorder (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 28 (30)
Cardiac failure acute (Cardiac disorders) | 19 (21)
Cardiac failure chronic (Cardiac disorders) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 183 (295)
Cardiac perforation (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 4 (4)
Cardiac valve disease (Cardiac disorders) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 20 (20)
Cardiogenic shock (Cardiac disorders) | 12 (12)
Cardiomyopathy (Cardiac disorders) | 18 (19)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 5 (5)
Cor pulmonale chronic (Cardiac disorders) | 1 (1)
Coronary artery aneurysm (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 120 (127)
Coronary artery dissection (Cardiac disorders) | 15 (15)
Coronary artery occlusion (Cardiac disorders) | 32 (32)
Coronary artery perforation (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 74 (76)
Coronary artery thrombosis (Cardiac disorders) | 9 (9)
Coronary ostial stenosis (Cardiac disorders) | 4 (4)
Electromechanical dissociation (Cardiac disorders) | 3 (3)
Extrasystoles (Cardiac disorders) | 1 (1)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 16 (16)
Left ventricular dysfunction (Cardiac disorders) | 5 (5)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 1 (1)
Mitral valve calcification (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 8 (9)
Mitral valve prolapse (Cardiac disorders) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 57 (59)
Myocardial ischaemia (Cardiac disorders) | 43 (44)
Palpitations (Cardiac disorders) | 11 (11)
Pericardial effusion (Cardiac disorders) | 5 (6)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 4 (4)
Pericarditis constrictive (Cardiac disorders) | 1 (1)
Post procedural myocardial infarction (Cardiac disorders) | 6 (6)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 23 (23)
Sinus arrest (Cardiac disorders) | 2 (2)
Sinus arrhythmia (Cardiac disorders) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sudden cardiac death (Cardiac disorders) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 11 (11)
Tachycardia (Cardiac disorders) | 2 (2)
Torsade de pointes (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 3 (3)
Ventricular asystole (Cardiac disorders) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 18 (18)
Ventricular flutter (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 40 (45)
Accidental death (General disorders) | 1 (1)
Adverse drug reaction (General disorders) | 4 (4)
Asthenia (General disorders) | 15 (15)
Catheter site haematoma (General disorders) | 21 (21)
Catheter site haemorrhage (General disorders) | 9 (9)
Chest pain (General disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Gait disturbance (General disorders) | 3 (3)
Generalised oedema (General disorders) | 2 (2)
Hernia (General disorders) | 1 (1)
Hernia obstructive (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Implant site discharge (General disorders) | 1 (1)
Infusion site phlebitis (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 10 (10)
Non-cardiac chest pain (General disorders) | 231 (311)
Oedema peripheral (General disorders) | 9 (9)
Organ failure (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 11 (13)
Sudden death (General disorders) | 3 (3)
Surgical failure (General disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 2 (2)
Unevaluable event (General disorders) | 1 (1)
Allergy to metals (Immune system disorders) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1)
Contrast media reaction (Immune system disorders) | 1 (1)
Dermatitis allergic (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 10 (10)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 2 (2)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 12 (12)
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 1 (1)
Device electrical finding (Injury, poisoning and procedural complications) | 3 (3)
Device lead damage (Injury, poisoning and procedural complications) | 1 (1)
Device malfunction (Injury, poisoning and procedural complications) | 2 (2)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1)
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 9 (10)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 160 (195)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (4)
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 1 (1)
Lead dislodgement (Injury, poisoning and procedural complications) | 1 (1)
Mechanical complication of implant (Injury, poisoning and procedural complications) | 2 (2)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Other injuries (Injury, poisoning and procedural complications) | 118 (139) — Other injuries consists of all the preferred terms which were not in Administration site reactions and Procedural and device related injuries high level group terms (HLGT) category for the corresponding system organ class (SOC).
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 (6)
Postoperative renal failure (Injury, poisoning and procedural complications) | 3 (3)
Procedural headache (Injury, poisoning and procedural complications) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 10 (10)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2)
Reperfusion injury (Injury, poisoning and procedural complications) | 7 (7)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Stent occlusion (Injury, poisoning and procedural complications) | 6 (6)
Stent-graft endoleak (Injury, poisoning and procedural complications) | 1 (2)
Thrombosis in device (Injury, poisoning and procedural complications) | 8 (9)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 2 (3)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 15 (15)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Others/Miscellaneous (Blood and lymphatic system disorders) | 89 (116)
Others/Miscellaneous (Congenital, familial and genetic disorders) | 10 (11)
Others/Miscellaneous (Ear and labyrinth disorders) | 3 (3)
Others/Miscellaneous (Endocrine disorders) | 5 (5)
Others/Miscellaneous (Eye disorders) | 10 (10)
Others/Miscellaneous (Gastrointestinal disorders) | 218 (277)
Others/Miscellaneous (Hepatobiliary disorders) | 55 (58)
Others/Miscellaneous (Infections and infestations) | 414 (585)
Others/Miscellaneous (Investigations) | 76 (83)
Others/Miscellaneous (Metabolism and nutrition disorders) | 106 (141)
Others/Miscellaneous (Musculoskeletal and connective tissue disorders) | 181 (194)
Others/Miscellaneous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 161 (184)
Others/Miscellaneous (Nervous system disorders) | 332 (386)
Others/Miscellaneous (Psychiatric disorders) | 42 (49)
Others/Miscellaneous (Reproductive system and breast disorders) | 12 (13)
Others/Miscellaneous (Respiratory, thoracic and mediastinal disorders) | 340 (485)
Others/Miscellaneous (Skin and subcutaneous tissue disorders) | 15 (15)
Others/Miscellaneous (Surgical and medical procedures) | 30 (30)
Other renal and urinary disorders (Renal and urinary disorders) | 95 (106) — Other renal and urinary disorders consist of all the preferred terms which were not in Acute renal failure for the corresponding system organ class.
Renal failure acute (Renal and urinary disorders) | 68 (72)
Accelerated hypertension (Vascular disorders) | 3 (3)
Aortic aneurysm (Vascular disorders) | 18 (19)
Aortic aneurysm rupture (Vascular disorders) | 3 (3)
Aortic dissection (Vascular disorders) | 2 (2)
Aortic intramural haematoma (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 4 (4)
Aorto-duodenal fistula (Vascular disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Arterial restenosis (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 2 (2)
Arterial thrombosis limb (Vascular disorders) | 2 (2)
Arteriosclerosis (Vascular disorders) | 19 (22)
Arteriovenous fistula (Vascular disorders) | 4 (5)
Arteriovenous malformation (Vascular disorders) | 1 (1)
Carotid arteriosclerosis (Vascular disorders) | 1 (1)
Carotid artery disease (Vascular disorders) | 7 (7)
Carotid artery occlusion (Vascular disorders) | 3 (3)
Carotid artery stenosis (Vascular disorders) | 46 (52)
Cerebral haemorrhage (Vascular disorders) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 24 (26)
Diverticulitis intestinal haemorrhagic (Vascular disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Vascular disorders) | 4 (4)
Duodenal ulcer haemorrhage (Vascular disorders) | 5 (5)
Embolism (Vascular disorders) | 1 (1)
Epistaxis (Vascular disorders) | 9 (9)
Femoral arterial stenosis (Vascular disorders) | 8 (9)
Femoral artery occlusion (Vascular disorders) | 7 (8)
Gastric haemorrhage (Vascular disorders) | 2 (2)
Gastric ulcer haemorrhage (Vascular disorders) | 7 (7)
Gastrointestinal haemorrhage (Vascular disorders) | 70 (77)
Gastrointestinal ulcer haemorrhage (Vascular disorders) | 3 (3)
Haemarthrosis (Vascular disorders) | 1 (1)
Haematemesis (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 4 (4)
Haemoptysis (Vascular disorders) | 5 (5)
Haemorrhage (Vascular disorders) | 1 (1)
Haemorrhage intracranial (Vascular disorders) | 8 (8)
Haemorrhagic erosive gastritis (Vascular disorders) | 2 (2)
Haemorrhagic stroke (Vascular disorders) | 2 (2)
Hepatic haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 24 (27)
Hypertensive crisis (Vascular disorders) | 7 (7)
Hypertensive emergency (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 33 (39)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 3 (3)
Iliac artery stenosis (Vascular disorders) | 3 (3)
Intermittent claudication (Vascular disorders) | 23 (29)
Ischaemic limb pain (Vascular disorders) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Vascular disorders) | 15 (15)
Mallory-Weiss syndrome (Vascular disorders) | 1 (1)
Mesenteric artery stenosis (Vascular disorders) | 2 (2)
Mesenteric occlusion (Vascular disorders) | 1 (1)
Oesophageal haemorrhage (Vascular disorders) | 1 (1)
Oesophageal varices haemorrhage (Vascular disorders) | 3 (3)
Operative haemorrhage (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 12 (14)
Pelvic haematoma (Vascular disorders) | 1 (1)
Peptic ulcer haemorrhage (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 10 (11)
Peripheral artery aneurysm (Vascular disorders) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 10 (12)
Peripheral vascular disorder (Vascular disorders) | 16 (19)
Petechiae (Vascular disorders) | 1 (1)
Pharyngeal haematoma (Vascular disorders) | 1 (1)
Portal vein thrombosis (Vascular disorders) | 1 (1)
Post procedural haematoma (Vascular disorders) | 1 (1)
Pulmonary artery thrombosis (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 15 (17)
Pulmonary hypertension (Vascular disorders) | 2 (2)
Renal artery occlusion (Vascular disorders) | 1 (1)
Renal artery stenosis (Vascular disorders) | 11 (11)
Renal hypertension (Vascular disorders) | 1 (1)
Retinal vascular occlusion (Vascular disorders) | 1 (1)
Retroperitoneal haematoma (Vascular disorders) | 2 (2)
Retroperitoneal haemorrhage (Vascular disorders) | 15 (15)
Skin ulcer (Vascular disorders) | 3 (3)
Subarachnoid haemorrhage (Vascular disorders) | 4 (4)
Subclavian artery stenosis (Vascular disorders) | 3 (3)
Subclavian steal syndrome (Vascular disorders) | 1 (1)
Subdural haematoma (Vascular disorders) | 13 (13)
Subdural haemorrhage (Vascular disorders) | 1 (1)
Superior vena caval occlusion (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4)
Ulcer haemorrhage (Vascular disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Vascular disorders) | 15 (15)
Vascular insufficiency (Vascular disorders) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 21 (21)
Vessel perforation (Vascular disorders) | 1 (1)
Wound haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XV-LTF Cohort (N=4852)
Angina pectoris (Cardiac disorders) | 644 (805)
Non-cardiac chest pain (General disorders) | 308 (366)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days